CLINICAL TRIAL: NCT00338130
Title: A Phase II, Multi-centre, Open-Label, Parallel Group, Randomised Study To Compare the Efficacy of AZD6244 vs Temozolomide in Patients With Unresectable AJCC Stage 3 or 4 Malignant Melanoma
Brief Title: Randomised Study to Compare the Efficacy of AZD6244 vs TMZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00003; EUDRACT No. 2006-001456-12
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Melanoma
Keywords: Melanoma; Phase II; AZD6244; temozolomide
MeSH Terms: conditions — Melanoma | interventions — AZD 6244; Temozolomide

ARMS (2):
- 1 (Active Comparator): Temozolomide
  Interventions: Drug: Temozolomide
- 2 (Experimental): AZD6244
  Interventions: Drug: AZD6244

INTERVENTIONS:
Drug: AZD6244 — Oral liquid or Capsule
  Other Names: ARRY-142886
  Arms: 2
Drug: Temozolomide — oral
  Arms: 1

SUMMARY:
The primary purpose of this study is to compare the efficacy of AZD6244 (ARRY-142886) with temozolomide in patients with advanced melanoma

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with late stage malignant melanoma
* Aged 18 or over
* Female patients must be post-menopausal or with negative urine pregnancy test if pre-menopausal

Exclusion Criteria:

* Any previous radiotherapy or chemotherapy (palliative radiotherapy is acceptable)
* Participation in any other trial with an investigational product within the previous 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of AZD6244 vs temozolomide in patients with unresectable AJCC stage 3 or 4 malignant melanoma by assessing progression free survival (PFS) | From date of randomisation until 6 months after first dose or study withdrawal (whichever is the earliest)
Time to death | From date of randomisation until 6 months after first dose or to date of death (whichever is the earliest)
Objective Response Rate | RECIST data collected as per institutional standard practise
Duration of response | RECIST data collected as per institutional standard practise

SECONDARY OUTCOMES:
Assessment of the safety and tolerability of AZD6244 | Assessed at all visits
Investigation of the pharmacokinetics of AZD6244 | Day 1 & 8 (for patients on AZD6244)
Assessment of the efficacy of AZD6244 versus temozolomide in patients who are BRAF and BRAF and /or NRAS mutation positive | From date of randomisation until 6 months after first dose or study withdrawal (whichever is the earliest)

CONTACTS AND LOCATIONS:
Overall Officials: AZD6244 Medical Science Director, MD, Study Director — AstraZeneca
Locations (33):
- United States (10):
  - Research Site, Santa Monica, California
  - Research Site, Aurora, Colorado
  - Research Site, Miami Beach, Florida
  - Research Site, Niles, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
- Argentina (2):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Vicente López
- Australia (3):
  - Research Site, Heidelberg
  - Research Site, Nedlands
  - Research Site, Waratah
- Austria (2):
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Oshawa, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Odense, Denmark
- France (3):
  - Research Site, Boulogne-Billancourt
  - Research Site, Nantes
  - Research Site, Villejuif
- Research Site, Zurich, Switzerland
- United Kingdom (3):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Oxford

REFERENCES:
- See also: CSR-1839IL-0151.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1530&filename=CSR-1839IL-0151.pdf